CLINICAL TRIAL: NCT00980005
Title: Immunogenicity & Safety Study of GSK Biologicals' Thimerosal-free Trivalent Influenza Vaccine (TIV) Versus a Licensed Comparator in Children
Brief Title: Study to Assess the Immunogenicity and Safety of an Investigational Influenza Vaccine in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 112999
Record Dates: First submitted 2009-09-17; First posted 2009-09-18 (Estimated); Results first posted 2012-02-15 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2016-09

CONDITIONS: Influenza
Keywords: GSK Biologicals influenza vaccine GSK1557482A; influenza infection
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Flulaval Group (Experimental): subjects received Flulaval™ vaccine according to their priming status and age:
  * 3-8 years: primed subjects 1 dose at Day 0; unprimed subjects 1 dose at Day 0 and a second dose at Day 28
  * 9-17 years: 1 dose at Day 0 Flulaval vaccine was administered intramuscularly into the non-dominant deltoid.
  Interventions: Biological: GSK investigational vaccine GSK1557482A
- Fluzone Group (Active Comparator): subjects received Fluzone® Sanofi Pasteur's vaccine according to their priming status and age:
  * 3-8 years: primed subjects 1 dose at Day 0; unprimed subjects 1 dose at Day 0 and a second dose at Day 28
  * 9-17 years: 1 dose at Day 0 Fluzone vaccine was administered intramuscularly into the non-dominant deltoid.
  Interventions: Biological: Fluzone®

INTERVENTIONS:
Biological: GSK investigational vaccine GSK1557482A — One intramuscular injection for primed subjects, two intramuscular injections for unprimed subjects
  Arms: Flulaval Group
Biological: Fluzone® — One intramuscular injection for primed subjects, two intramuscular injections for unprimed subjects
  Arms: Fluzone Group

SUMMARY:
The objective of this study is to evaluate the immunogenicity and safety of GSK Biologicals' investigational vaccine GSK1557482A.

ELIGIBILITY:
Inclusion Criteria:

* Subjects and/or subject parent(s)/Legally Acceptable Representative(s) (LAR) who the investigator believes can and will comply with the requirements of the protocol.
* A male or female child aged between 3 years and 17 years of age at the time of the first vaccination; children who may or may not have had previous administration of influenza vaccine in a previous season are acceptable.
* Written informed consent obtained from the subject/from the parent(s)/LAR(s) of the subject.
* Healthy subjects as established by medical history and history-directed clinical examination before entering into the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:
* has practiced adequate contraception for 30 days prior to vaccination, and
* has a negative pregnancy test on the day of vaccination, and
* has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the administration of the study vaccine, or planned use during the study period. Routine, registered childhood vaccinations or registered and recommended pandemic influenza vaccine are not an exclusion.
* Receipt of a seasonal influenza vaccine outside of this study, during current (2009-2010) flu season.
* Child in care
* Receipt of systemic glucocorticoids within 1 month prior to study enrollment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrollment. Topical, intra-articular or inhaled glucocorticoids are allowed.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* History of hypersensitivity to any vaccine.
* History of Guillain-Barré-syndrome within 6 weeks of receipt of prior inactivated influenza virus vaccine.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine(s).
* Acute disease and/or fever at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2116 (Actual)
Dates: Start 2009-10-13; Primary Completion 2010-03-02 (Actual); Study Completion 2010-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (28):
- United States (28):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Benton, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Woodstock, Georgia
  - GSK Investigational Site, DeKalb, Illinois
  - GSK Investigational Site, Newton, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Woburn, Massachusetts
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Cortland, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Austintown, Ohio
  - GSK Investigational Site, Albany, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Orem, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Burke, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Li-Kim-Moy J, Wood N, Jones C, Macartney K, Booy R. Impact of Fever and Antipyretic Use on Influenza Vaccine Immune Reponses in Children. Pediatr Infect Dis J. 2018 Oct;37(10):971-975. doi: 10.1097/INF.0000000000001949. PMID 29465480
- [Derived] Domachowske JB, Blatter M, Chandrasekaran V, Liu A, Jain VK, Fries L. A randomized, controlled trial in children to assess the immunogenicity and safety of a thimerosal-free trivalent seasonal influenza vaccine. Pediatr Infect Dis J. 2012 Jun;31(6):605-15. doi: 10.1097/INF.0b013e31824e2924. PMID 22333695
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 112999 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112999 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112999 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112999 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112999 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112999 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112999 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were stratified by age-strata: 3-4, 5-8 and 9-17 years and received vaccine according to their priming status: primed subjects received a 2-dose priming immunization in a previous season, whereas unprimed subjects had not. Blood samples: at Days 0 - 28 for primed subjects and subjects 9-17 years and at Days 0-56 for unprimed subjects.
Period: Overall Study
Arm/Group | Flulaval Group | Fluzone Group
Started | 1055 | 1061
Completed | 1008 | 998
Not Completed | 47 | 63
Not completed — Withdrawal by Subject | 6 | 17
Not completed — Lost to Follow-up | 37 | 43
Not completed — Other | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flulaval Group | Fluzone Group | Total
Number analyzed (Participants) | 1055 | 1061 | 2116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.8 (4.18) | 7.8 (4.10) | 7.8 (4.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 500 | 496 | 996
  Male | 555 | 565 | 1120

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean of Haemagglutination Inhibiting (HI) Antibodies Titers Against the Three Strains.
Description: The three strains assessed were A/Brisbane/59/2007 (H1N1), A/Uruguay/716/2007 (H3N2) and B/Brisbane/60/2008.
  Titers were expressed as geometric mean antibody titers (GMTs).
Time Frame: At Day 0 and 28 after last vaccine dose.
Population: The According-To-Protocol cohort for immunogenicity included all evaluable subjects for whom data concerning immunogenicity outcome measures were available. This included subjects for whom assay results were available for antibodies against at least one vaccine strain after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 987 | 979
Titers
  A/Brisbane [at Day 0]: number analyzed (Participants) | 987 | 978
  A/Brisbane [at Day 0] | 46.0 [41.9 to 50.4] | 45.8 [41.8 to 50.2]
  A/Brisbane [at Day 28] | 320.9 [298.3 to 345.2] | 329.4 [306.8 to 353.7]
  A/Uruguay [at Day 0]: number analyzed (Participants) | 987 | 978
  A/Uruguay [at Day 0] | 57.1 [51.8 to 63.0] | 63.9 [58.1 to 70.3]
  A/Uruguay [at Day 28] | 414.7 [386.5 to 444.9] | 451.9 [423.8 to 481.8]
  B/Brisbane [at Day 0]: number analyzed (Participants) | 987 | 978
  B/Brisbane [at Day 0] | 16.6 [15.3 to 18.1] | 16.8 [15.4 to 18.3]
  B/Brisbane [at Day 28] | 213.7 [198.5 to 230.1] | 200.2 [186.1 to 215.3]

2. Primary Outcome: Number of Seroconverted Subjects for HI Antibodies Against the Three Strains.
Description: The three strains assessed were A/Brisbane/59/2007 (H1N1), A/Uruguay/716/2007 (H3N2) and B/Brisbane/60/2008.
  Seroconversion was defined as the percentage of vaccinees that had either a pre-vaccination (Day 0) titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-vaccination titer.
Time Frame: At Day 28 after last vaccine dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 987 | 978
Participants
  A/Brisbane | 590 | 569
  A/Uruguay | 673 | 647
  B/Brisbane | 800 | 769

3. Secondary Outcome: Geometric Mean of Haemagglutination Inhibiting (HI) Antibodies Titers Against the Three Strains, by Age-strata.
Description: The three strains assessed were A/Brisbane/59/2007 (H1N1), A/Uruguay/716/2007 (H3N2) and B/Brisbane/60/2008.
  Titers were expressed as geometric mean antibody titers (GMTs).
  Subjects in each group were also stratified in the following age-strata: 3-4 years, 5-8 years and 9-17 years.
Time Frame: At Day 0 and 28 after last vaccine dose.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 987 | 979
Titers
  A/Brisbane at Day 0 [3-4 years]: number analyzed (Participants) | 275 | 260
  A/Brisbane at Day 0 [3-4 years] | 38.4 [31.5 to 46.7] | 34.4 [28.4 to 41.7]
  A/Brisbane at Day 28 [3-4 years]: number analyzed (Participants) | 275 | 260
  A/Brisbane at Day 28 [3-4 years] | 263.5 [229.3 to 302.9] | 281.9 [246.3 to 322.7]
  A/Brisbane at Day 0 [5-8 years]: number analyzed (Participants) | 353 | 353
  A/Brisbane at Day 0 [5-8 years] | 40.2 [34.8 to 46.5] | 41.4 [35.7 to 48.1]
  A/Brisbane at Day 28 [5-8 years]: number analyzed (Participants) | 353 | 354
  A/Brisbane at Day 28 [5-8 years] | 251.8 [222.3 to 285.3] | 251.5 [223.8 to 282.7]
  A/Brisbane at Day 0 [9-17 years]: number analyzed (Participants) | 359 | 365
  A/Brisbane at Day 0 [9-17 years] | 60.2 [52.0 to 69.6] | 61.9 [53.7 to 71.2]
  A/Brisbane at Day 28 [9-17 years]: number analyzed (Participants) | 359 | 365
  A/Brisbane at Day 28 [9-17 years] | 473.6 [425.1 to 527.5] | 478.2 [428.2 to 534.0]
  A/Uruguay at Day 0 [3-4 years]: number analyzed (Participants) | 275 | 260
  A/Uruguay at Day 0 [3-4 years] | 38.7 [31.7 to 47.2] | 50.2 [40.7 to 61.8]
  A/Uruguay at Day 28 [3-4 years]: number analyzed (Participants) | 275 | 260
  A/Uruguay at Day 28 [3-4 years] | 322.8 [276.9 to 376.3] | 418.3 [366.9 to 477.0]
  A/Uruguay at Day 0 [5-8 years]: number analyzed (Participants) | 353 | 353
  A/Uruguay at Day 0 [5-8 years] | 78.5 [66.9 to 92.1] | 78.1 [67.0 to 91.2]
  A/Uruguay at Day 28 [5-8 years]: number analyzed (Participants) | 353 | 354
  A/Uruguay at Day 28 [5-8 years] | 476.3 [426.3 to 532.1] | 494.2 [442.4 to 552.1]
  A/Uruguay at Day 0 [9-17 years]: number analyzed (Participants) | 359 | 365
  A/Uruguay at Day 0 [9-17 years] | 56.3 [48.7 to 65.2] | 62.6 [54.1 to 72.3]
  A/Uruguay at Day 28 [9-17 years]: number analyzed (Participants) | 359 | 365
  A/Uruguay at Day 28 [9-17 years] | 438.4 [394.1 to 487.6] | 437.8 [397.4 to 482.3]
  B/Brisbane at Day 0 [3-4 years]: number analyzed (Participants) | 275 | 260
  B/Brisbane at Day 0 [3-4 years] | 13.1 [11.2 to 15.3] | 11.6 [10.0 to 13.5]
  B/Brisbane at Day 28 [3-4 years]: number analyzed (Participants) | 275 | 260
  B/Brisbane at Day 28 [3-4 years] | 174.1 [149.8 to 202.5] | 148.5 [129.4 to 170.4]
  B/Brisbane at Day 0 [5-8 years]: number analyzed (Participants) | 353 | 353
  B/Brisbane at Day 0 [5-8 years] | 16.2 [14.1 to 18.7] | 16.9 [14.7 to 19.5]
  B/Brisbane at Day 28 [5-8 years]: number analyzed (Participants) | 353 | 354
  B/Brisbane at Day 28 [5-8 years] | 196.8 [175.1 to 221.1] | 202.8 [179.0 to 229.7]
  B/Brisbane at Day 0 [9-17 years]: number analyzed (Participants) | 359 | 365
  B/Brisbane at Day 0 [9-17 years] | 20.5 [17.9 to 23.6] | 21.7 [18.9 to 24.9]
  B/Brisbane at Day 28 [9-17 years]: number analyzed (Participants) | 359 | 365
  B/Brisbane at Day 28 [9-17 years] | 271.1 [240.8 to 305.1] | 244.6 [217.9 to 274.5]

4. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Titers Against the Three Strains, by Age-strata.
Description: The three strains assessed were A/Brisbane/59/2007 (H1N1), A/Uruguay/716/2007 (H3N2) and B/Brisbane/60/2008.
  Seroconversion was defined as the percentage of vaccinees that had either a pre-vaccination (Day 0) titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a four-fold increase in post-vaccination titer.
  Subjects in each group were also stratified in the following age-strata: 3-4 years, 5-8 years and 9-17 years.
Time Frame: At Day 28 after last vaccine dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 987 | 978
Participants
  A/Brisbane [3-4 years]: number analyzed (Participants) | 275 | 260
  A/Brisbane [3-4 years] | 161 | 177
  A/Brisbane [5-8 years]: number analyzed (Participants) | 353 | 353
  A/Brisbane [5-8 years] | 211 | 191
  A/Brisbane [9-17 years]: number analyzed (Participants) | 359 | 365
  A/Brisbane [9-17 years] | 218 | 201
  A/Uruguay [3-4 years]: number analyzed (Participants) | 275 | 260
  A/Uruguay [3-4 years] | 203 | 190
  A/Uruguay [5-8 years]: number analyzed (Participants) | 353 | 353
  A/Uruguay [5-8 years] | 233 | 228
  A/Uruguay [9-17 years]: number analyzed (Participants) | 359 | 365
  A/Uruguay [9-17 years] | 237 | 229
  B/Brisbane [3-4 years]: number analyzed (Participants) | 275 | 260
  B/Brisbane [3-4 years] | 227 | 214
  B/Brisbane [5-8 years]: number analyzed (Participants) | 353 | 353
  B/Brisbane [5-8 years] | 289 | 293
  B/Brisbane [9-17 years]: number analyzed (Participants) | 359 | 365
  B/Brisbane [9-17 years] | 284 | 262

5. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies Titers Against the Three Strains.
Description: The three strains assessed were A/Brisbane/59/2007 (H1N1), A/Uruguay/716/2007 (H3N2) and B/Brisbane/60/2008.
  Seroprotection rate (SPR) was defined as the percentage of vaccinees with a serum HI titer ≥ 1:40 that represents a putative protective level in adults.
Time Frame: At Day 0 and 28 after last vaccine dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 987 | 979
Participants
  A/Brisbane [at Day 0]: number analyzed (Participants) | 987 | 978
  A/Brisbane [at Day 0] | 640 | 639
  A/Brisbane [at Day 28] | 969 | 965
  A/Uruguay [at Day 0]: number analyzed (Participants) | 987 | 978
  A/Uruguay [at Day 0] | 676 | 690
  A/Uruguay [at Day 28] | 970 | 973
  B/Brisbane [at Day 0]: number analyzed (Participants) | 987 | 978
  B/Brisbane [at Day 0] | 359 | 360
  B/Brisbane [at Day 28] | 936 | 925

6. Secondary Outcome: Number of Seroprotected Subjects for HI Antibodies Titers Against the Three Strains, by Age-strata.
Description: The three strains assessed were A/Brisbane/59/2007 (H1N1), A/Uruguay/716/2007 (H3N2) and B/Brisbane/60/2008.
  Seroprotection rate (SPR) was defined as the percentage of vaccinees with a serum HI titer ≥ 1:40 that represents a putative protective level in adults.
  Subjects in each group were also stratified in the following age-strata: 3-4 years, 5-8 years and 9-17 years.
Time Frame: At Day 0 and 28 after last vaccine dose.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 987 | 979
Participants
  A/Brisbane at Day 0 [3-4 years]: number analyzed (Participants) | 275 | 260
  A/Brisbane at Day 0 [3-4 years] | 155 | 145
  A/Brisbane at Day 28 [3-4 years]: number analyzed (Participants) | 275 | 260
  A/Brisbane at Day 28 [3-4 years] | 265 | 258
  A/Brisbane at Day 0 [5-8 years]: number analyzed (Participants) | 353 | 353
  A/Brisbane at Day 0 [5-8 years] | 227 | 228
  A/Brisbane at Day 28 [5-8 years]: number analyzed (Participants) | 353 | 354
  A/Brisbane at Day 28 [5-8 years] | 347 | 346
  A/Brisbane at Day 0 [9-17 years]: number analyzed (Participants) | 359 | 365
  A/Brisbane at Day 0 [9-17 years] | 258 | 266
  A/Brisbane at Day 28 [9-17 years]: number analyzed (Participants) | 359 | 365
  A/Brisbane at Day 28 [9-17 years] | 357 | 361
  A/Uruguay at Day 0 [3-4 years]: number analyzed (Participants) | 275 | 260
  A/Uruguay at Day 0 [3-4 years] | 153 | 158
  A/Uruguay at Day 28 [3-4 years]: number analyzed (Participants) | 275 | 260
  A/Uruguay at Day 28 [3-4 years] | 265 | 259
  A/Uruguay at Day 0 [5-8 years]: number analyzed (Participants) | 353 | 353
  A/Uruguay at Day 0 [5-8 years] | 267 | 269
  A/Uruguay at Day 28 [5-8 years]: number analyzed (Participants) | 353 | 354
  A/Uruguay at Day 28 [5-8 years] | 349 | 351
  A/Uruguay at Day 0 [9-17 years]: number analyzed (Participants) | 359 | 365
  A/Uruguay at Day 0 [9-17 years] | 256 | 263
  A/Uruguay at Day 28 [9-17 years] ): number analyzed (Participants) | 359 | 365
  A/Uruguay at Day 28 [9-17 years] ) | 356 | 363
  B/Brisbane at Day 0 [3-4 years]: number analyzed (Participants) | 275 | 260
  B/Brisbane at Day 0 [3-4 years] | 80 | 68
  B/Brisbane at Day 28 [3-4 years]: number analyzed (Participants) | 275 | 260
  B/Brisbane at Day 28 [3-4 years] | 254 | 239
  B/Brisbane at Day 0 [5-8 years]: number analyzed (Participants) | 353 | 353
  B/Brisbane at Day 0 [5-8 years] | 127 | 127
  B/Brisbane at Day 28 [5-8 years]: number analyzed (Participants) | 353 | 354
  B/Brisbane at Day 28 [5-8 years] | 334 | 335
  B/Brisbane at Day 0 [9-17 years]: number analyzed (Participants) | 359 | 365
  B/Brisbane at Day 0 [9-17 years] | 152 | 165
  B/Brisbane at Day 28 [9-17 years]: number analyzed (Participants) | 359 | 365
  B/Brisbane at Day 28 [9-17 years] | 348 | 351

7. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Titers Against the Three Strains.
Description: The three strains assessed were A/Brisbane/59/2007 (H1N1), A/Uruguay/716/2007 (H3N2) and B/Brisbane/60/2008.
  Seroconversion factor (SCF) was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination.
  Seroconversion factor (SCF) was defined as the geometric mean of the within subjects ratios of the post-vaccination reciprocal HI titer to the Day 0 reciprocal HI titer. SCFs were calculated at Day 28 following the complete vaccination regimen.
Time Frame: At Day 0 and at Day 28 after last vaccine dose
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 987 | 978
Fold change
  A/Brisbane | 7.0 [6.3 to 7.7] | 7.2 [6.5 to 8.0]
  A/Uruguay | 7.3 [6.7 to 7.9] | 7.1 [6.5 to 7.7]
  B/Brisbane | 12.8 [11.8 to 14.0] | 11.9 [10.9 to 13.0]

8. Secondary Outcome: Seroconversion Factor (SCF) for HI Antibodies Titers Against the Three Strains, by Age-strata.
Description: The three strains assessed were A/Brisbane/59/2007 (H1N1), A/Uruguay/716/2007 (H3N2) and B/Brisbane/60/2008.
  Seroconversion factor (SCF) was defined as the fold increase in serum HI GMTs post-vaccination compared to pre-vaccination.
  Seroconversion factor (SCF) was defined as the geometric mean of the within subjects ratios of the post-vaccination reciprocal HI titer to the Day 0 reciprocal HI titer. SCFs were calculated at Day 28 following the complete vaccination regimen.
  Subjects in each group were also stratified in the following age-strata: 3-4 years, 5-8 years and 9-17 years.
Time Frame: At Day 0 and at Day 28 after last vaccine dose
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Fold change
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 987 | 978
Fold change
  A/Brisbane [3-4 years]: number analyzed (Participants) | 275 | 260
  A/Brisbane [3-4 years] | 6.9 [5.7 to 8.2] | 8.2 [6.8 to 9.8]
  A/Brisbane [5-8 years]: number analyzed (Participants) | 353 | 353
  A/Brisbane [5-8 years] | 6.3 [5.4 to 7.3] | 6.1 [5.2 to 7.1]
  A/Brisbane [9-17 years]: number analyzed (Participants) | 359 | 365
  A/Brisbane [9-17 years] | 7.9 [6.7 to 9.3] | 7.7 [6.5 to 9.2]
  A/Uruguay [3-4 years]: number analyzed (Participants) | 275 | 260
  A/Uruguay [3-4 years] | 8.4 [7.2 to 9.7] | 8.3 [7.1 to 9.9]
  A/Uruguay [5-8 years]: number analyzed (Participants) | 353 | 353
  A/Uruguay [5-8 years] | 6.1 [5.3 to 6.9] | 6.3 [5.5 to 7.2]
  A/Uruguay [9-17 years]: number analyzed (Participants) | 359 | 365
  A/Uruguay [9-17 years] | 7.8 [6.7 to 9.0] | 7.0 [6.0 to 8.2]
  B/Brisbane [3-4 years]: number analyzed (Participants) | 275 | 260
  B/Brisbane [3-4 years] | 13.3 [11.5 to 15.4] | 12.8 [11.0 to 14.8]
  B/Brisbane [5-8 years]: number analyzed (Participants) | 353 | 353
  B/Brisbane [5-8 years] | 12.2 [10.7 to 13.8] | 12.0 [10.5 to 13.7]
  B/Brisbane [9-17 years]: number analyzed (Participants) | 359 | 365
  B/Brisbane [9-17 years] | 13.2 [11.3 to 15.4] | 11.3 [9.6 to 13.2]

9. Secondary Outcome: Number of Subjects Below 5 Years of Age With Any, Severe (Grade 3) and Related to Vaccination Solicited General Adverse Events (AEs).
Description: The general symptoms solicited from study subjects younger than 5 years of age were drowsiness, irritability, loss of appetite, and fever(= axillary temperature equal to or above 38.0 degrees Celsius (°C)).
  Any = occurrence of any solicited general symptom regardless of intensity grade or relationship to vaccination.
  Grade 3 drowsiness, irritability = symptom that prevented normal activity. Grade 3 loss of appetite = not eating at all.
  Grade 3 temperature = axillary temperature ≥ 39.0°C and ≤ 40.0°C.
  Related = symptom assessed by the investigator as causally related to the vaccination.
Time Frame: During a 4-day follow-up period (Days 0-3) after vaccination.
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Flulaval Less Than 5 Years Old Group: Subjects below 5 years of age and who received 1 or 2 injections of Flulaval™ vaccine according to their priming status.
- Fluzone Les Than 5 Years Old Group: Subjects below 5 years of age and who received 1 or 2 injections of Fluzone® Sanofi Pasteur's vaccine according to their priming status and age
Arm/Group | Flulaval Group | Fluzone Group | Flulaval Less Than 5 Years Old Group | Fluzone Les Than 5 Years Old Group
Number analyzed (Participants) | 0 | 0 | 293 | 279
Participants
  Any drowsiness |  |  | 61 | 63
  Grade 3 drowsiness |  |  | 4 | 2
  Drowsiness related to vaccination |  |  | 57 | 56
  Any irritability |  |  | 86 | 87
  Grade 3 irritability |  |  | 6 | 4
  Irritability related to vaccination |  |  | 81 | 81
  Any loss of appetite |  |  | 52 | 47
  Grade 3 loss of appetite |  |  | 7 | 2
  Loss of appetite related to vaccination |  |  | 45 | 42
  Fever >= 38.0°C |  |  | 15 | 10
  Fever >= 39.0°C - <= 40.0°C |  |  | 3 | 2
  Fever related to vaccination |  |  | 14 | 8

10. Secondary Outcome: Number of Subjects of 5 Years of Age and Above Reporting Any, Severe (Grade 3) and Related to Vaccination Solicited General Adverse Events (AEs).
Description: The general symptoms solicited from study subjects 5 years of age and older were arthralgia (joint pain), fatigue, headache, muscle aches, shivering, and fever(= axillary temperature equal to or above 38.0 degrees Celsius (°C)).
  Any = occurrence of any solicited general symptom regardless of intensity grade or relationship to vaccination.
  Grade 3 symptoms = symptoms that prevented normal activity. Grade 3 temperature = axillary temperature ≥ 39.0°C and ≤ 40.0°C.
  Related = symptom assessed by the investigator as causaly related to the vaccination.
Time Frame: During a 4-day follow-up period (Days 0-3) after vaccination.
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Groups:
- Flulaval 5 Years of Age and Older Group: Subjects aged 5 years and above and who received 1 or 2 injections of Flulaval™ vaccine according to their priming status.
- Fluzone 5 Years of Age and Older Group: Subjects aged 5 years and above and who received 1 or 2 injections of Fluzone® Sanofi Pasteur's vaccine according to their priming status and age
Arm/Group | Flulaval Group | Fluzone Group | Flulaval 5 Years of Age and Older Group | Fluzone 5 Years of Age and Older Group
Number analyzed (Participants) | 0 | 0 | 750 | 747
Participants
  Any arthralgia |  |  | 70 | 80
  Grade 3 arthralgia |  |  | 2 | 2
  Arthralgia related to vaccination |  |  | 65 | 74
  Any fatigue |  |  | 138 | 137
  Grade 3 fatigue |  |  | 11 | 10
  Fatigue related to vaccination |  |  | 119 | 117
  Any headache |  |  | 141 | 131
  Grade 3 headache |  |  | 6 | 4
  Headache related to vaccination |  |  | 115 | 105
  Any muscle aches |  |  | 200 | 189
  Grade 3 muscle aches |  |  | 6 | 7
  Muscle aches related to vaccination |  |  | 180 | 179
  Any shivering |  |  | 45 | 40
  Grade 3 shivering |  |  | 2 | 3
  Shivering related to vaccination |  |  | 36 | 31
  Fever >= 38.0°C |  |  | 36 | 36
  Fever >= 39.0°C - <= 40.0°C |  |  | 12 | 13
  Temperature related to vaccination |  |  | 27 | 25

11. Secondary Outcome: Number of Subjects Reporting Any and Severe (Grade 3) Solicited Local Adverse Events (AEs).
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of any solicited general symptom regardless of intensity grade.
  Grade 3 pain = pain that prevented normal activity. Grade 3 redness, swelling = redness, swelling above 100 millimeter (mm). All solicited local AEs were considered to be causally related to vaccination.
Time Frame: During a 4-day follow-up period (Days 0-3) after vaccination.
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 1043 | 1026
Participants
  Any pain | 615 | 584
  Grade 3 pain | 26 | 28
  Any redness | 57 | 53
  Grade 3 redness | 2 | 1
  Any swelling | 51 | 59
  Grade 3 swelling | 1 | 0

12. Secondary Outcome: Number of Subjects Reporting Any and Severe (Grade 3) Solicited Local Adverse Events (AEs), by Age-strata.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = occurrence of any solicited general symptom regardless of intensity grade.
  Grade 3 pain = pain that prevented normal activity. Grade 3 redness, swelling = redness, swelling above 100 millimeter (mm). All solicited local AEs were considered to be causally related to vaccination. Subjects in each group were also stratified in the following age-strata: 3-4 years, 5-8 years and 9-17 years.
Time Frame: During a 4-day follow-up period (Days 0-3) after vaccination.
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 1043 | 1026
Participants
  Any pain [3-4 years]: number analyzed (Participants) | 294 | 281
  Any pain [3-4 years] | 139 | 130
  Grade 3 pain [3-4 years]: number analyzed (Participants) | 294 | 281
  Grade 3 pain [3-4 years] | 5 | 4
  Any redness [3-4 years]: number analyzed (Participants) | 294 | 281
  Any redness [3-4 years] | 14 | 18
  Grade 3 redness [3-4 years]: number analyzed (Participants) | 294 | 281
  Grade 3 redness [3-4 years] | 0 | 0
  Any swelling [3-4 years]: number analyzed (Participants) | 294 | 281
  Any swelling [3-4 years] | 9 | 11
  Grade 3 swelling [3-4 years]: number analyzed (Participants) | 294 | 281
  Grade 3 swelling [3-4 years] | 0 | 0
  Any pain [5-8 years]: number analyzed (Participants) | 387 | 377
  Any pain [5-8 years] | 252 | 249
  Grade 3 pain [5-8 years]: number analyzed (Participants) | 387 | 377
  Grade 3 pain [5-8 years] | 16 | 18
  Any redness [5-8 years]: number analyzed (Participants) | 387 | 377
  Any redness [5-8 years] | 30 | 22
  Grade 3 redness [5-8 years]: number analyzed (Participants) | 387 | 377
  Grade 3 redness [5-8 years] | 2 | 1
  Any swelling [5-8 years]: number analyzed (Participants) | 387 | 377
  Any swelling [5-8 years] | 24 | 28
  Grade 3 swelling [5-8 years]: number analyzed (Participants) | 387 | 377
  Grade 3 swelling [5-8 years] | 1 | 0
  Any pain [9-17 years]: number analyzed (Participants) | 362 | 368
  Any pain [9-17 years] | 224 | 205
  Grade 3 pain [9-17 years]: number analyzed (Participants) | 362 | 368
  Grade 3 pain [9-17 years] | 5 | 6
  Any redness [9-17 years]: number analyzed (Participants) | 362 | 368
  Any redness [9-17 years] | 13 | 13
  Grade 3 redness [9-17 years]: number analyzed (Participants) | 362 | 368
  Grade 3 redness [9-17 years] | 0 | 0
  Any swelling [9-17 years]: number analyzed (Participants) | 362 | 368
  Any swelling [9-17 years] | 18 | 20
  Grade 3 swelling [9-17 years]: number analyzed (Participants) | 362 | 368
  Grade 3 swelling [9-17 years] | 0 | 0

13. Secondary Outcome: Number of Subjects Reporting Any, Severe (Grade 3) and Related to Vaccination Unsolicited Adverse Events (AEs).
Description: Any adverse event (AE) reported in addition to those solicited during the clinical study. Also any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
  Grade 3 = event that prevented normal activities. Related = event assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 28 day follow-up period (Days 0-27) after vaccination.
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 1055 | 1061
Participants
  Any AE(s) | 421 | 387
  Grade 3 AE(s) | 81 | 83
  Related AE(s) | 65 | 57

14. Secondary Outcome: Number of Subjects Reporting Any, Severe (Grade 3) and Related to Vaccination Unsolicited Adverse Events (AEs), by Age-strata.
Description: Any adverse event (AE) reported in addition to those solicited during the clinical study. Also any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
  Subjects in each group were also stratified in the following age-strata: 3-4 years, 5-8 years and 9-17 years.
  Grade 3 = event that prevented normal activities. Related = event assessed by the investigator as causally related to the study vaccination.
Time Frame: During a 28 day follow-up period (Days 0-27) after vaccination.
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 1055 | 1061
Participants
  Any AE(s) [3-4 years]: number analyzed (Participants) | 298 | 295
  Any AE(s) [3-4 years] | 134 | 128
  Grade 3 AE(s) [3-4 years]: number analyzed (Participants) | 298 | 295
  Grade 3 AE(s) [3-4 years] | 23 | 25
  Related AE(s) [3-4 years]: number analyzed (Participants) | 298 | 295
  Related AE(s) [3-4 years] | 17 | 16
  Any AE(s) [5-8 years]: number analyzed (Participants) | 390 | 393
  Any AE(s) [5-8 years] | 175 | 149
  Grade 3 AE(s) [5-8 years]: number analyzed (Participants) | 390 | 393
  Grade 3 AE(s) [5-8 years] | 36 | 32
  Related AE(s) [5-8 years]: number analyzed (Participants) | 390 | 393
  Related AE(s) [5-8 years] | 32 | 24
  Any AE(s) [9-17 years]: number analyzed (Participants) | 367 | 373
  Any AE(s) [9-17 years] | 112 | 110
  Grade 3 AE(s) [9-17 years]: number analyzed (Participants) | 367 | 373
  Grade 3 AE(s) [9-17 years] | 22 | 26
  Related AE(s) [9-17 years]: number analyzed (Participants) | 367 | 373
  Related AE(s) [9-17 years] | 16 | 17

15. Secondary Outcome: Number of Subjects Reporting Medically Attended Adverse Events (MAEs).
Description: For each solicited and unsolicited symptom the subject experiences, the subject/subject's parent(s)/ Legally Acceptable Representative (LAR(s)) was asked if they received medical attention defined as hospitalisation, an emergency room visit or a visit to or from medical personnel (medical doctor) for any reason.
Time Frame: During the entire study period (From Day 0 up to Day 180).
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 1055 | 1061
Participants | 447 | 432

16. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs).
Description: An SAE is defined as any untoward medical occurrence in a patient or clinical investigation subject that: results in death, is lifethreatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.
Time Frame: During the entire study period (From Day 0 up to Day 180).
Population: The Total Vaccinated cohort included all vaccinated subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Flulaval Group | Fluzone Group
Number analyzed (Participants) | 1055 | 1061
Participants | 10 | 6

ADVERSE EVENTS:
Time Frame: Solicited AEs: During a 4-day follow-up period (Days 0-3) after vaccination; Unsolicited AEs:During a 28 day follow-up period (Days 0-27) after vaccination.; SAEs: During the entire study period (From Day 0 up to Day 180).
Description: Safety data were collected and tabulated for all subjects regardless of age categories but solicited general symptoms were collected and tabulated for subjects below 5 years of age and for subjects of 5 years of age and above. Solicited symtoms were assessed for subjects who daily recorded AEs and who returned the diary card post-vaccination.
Arm/Group | Flulaval Group | Fluzone Group
Serious Adverse Events (participants affected / at risk) | 10/1055 | 6/1061
Other Adverse Events (participants affected / at risk) | 742/1055 | 710/1061
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flulaval Group (N=1055) | Fluzone Group (N=1061)
Pneumonia (Infections and infestations) | 2 | 1
Herpangina (Infections and infestations) | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 1 | 0
Affective disorder (Psychiatric disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
H1N1 influenza (Infections and infestations) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oppositional defiant disorder (Psychiatric disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Type 1 diabetes mellitus (Immune system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Flulaval Group (N=1055) | Fluzone Group (N=1061)
Cough (Respiratory, thoracic and mediastinal disorders) | 129 | 115 — Unsolicited AE
Pyrexia (General disorders) | 62 | 60 — Unsolicited AE
Arthralgia (General disorders) | 70/750 | 80/747 — Solicited general AE: Subjects of 5 years of age and above
Fatigue (General disorders) | 138/750 | 137/747 — Solicited general AE: Subjects of 5 years of age and above
Headache (General disorders) | 141/750 | 131/747 — Solicited general AE: Subjects of 5 years of age and above
Muscle aches (General disorders) | 200/750 | 189/747 — Solicited general AE: Subjects of 5 years of age and above
Shivering (General disorders) | 45/750 | 40/747 — Solicited general AE: Subjects of 5 years of age and above
Drowsiness (General disorders) | 61/293 | 63/279 — Solicited general AE: Subjects below 5 years of age
Irritability (General disorders) | 86/293 | 87/279 — Solicited general AE: Subjects below 5 years of age
Loss of appetite (General disorders) | 52/293 | 47/279 — Solicited general AE: Subjects below 5 years of age
Temperature (General disorders) | 15/293 | 10/279 — Solicited general AE: Subjects below 5 years of age. Temperature = axillary temperature equal to or above 38.0 degrees Celsius (°C).
Pain (General disorders) | 615/1043 | 584/1026 — Solicited local AE
Redness (General disorders) | 57/1043 | 53/1026 — Solicited local AE
Swelling (General disorders) | 51/1043 | 59/1026 — Solicited local AE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.